CLINICAL TRIAL: NCT00092079
Title: A 15-Week, Double-Blind, Randomized, Active-Controlled, Multi-Center Study With 24-Week Extension to Evaluate the Safety, Tolerability, Efficacy of Alendronate 70 mg Plus Vitamin D3 2800 IU Combination Tablet in Men and Postmenopausal Women With Osteoporosis
Brief Title: A Study of MK0217A and Dietary Supplement in Men and Postmenopausal Women With Osteoporosis (0217A-227)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217A-227 Extension; 2004_021
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Osteoporosis; Vitamin D Deficiency
MeSH Terms: conditions — Osteoporosis; Vitamin D Deficiency | interventions — Alendronate; Cholecalciferol; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217A, alendronate sodium (+) cholecalciferol / Duration of Treatment: 24 weeks

SUMMARY:
The purpose of this study is to test the safety, tolerability, and effectiveness of an investigational drug and dietary supplement to reduce the risk of vitamin D insufficiency and deficiency during treatment of osteoporosis in men and postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal women who are osteoporotic

Exclusion Criteria:

* Vitamin D deficiency
* Other disease of bone or mineral metabolism
* Digestive disease causing malabsorption
* Other medical conditions that are not adequately treated

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2004-01; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability; primary parameter assessed is the proportion of patients who develop hypercalcuria

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitior, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Recker R, Lips P, Felsenberg D, Lippuner K, Benhamou L, Hawkins F, Delmas PD, Rosen C, Emkey R, Salzmann G, He W, Santora AC. Alendronate with and without cholecalciferol for osteoporosis: results of a 15-week randomized controlled trial. Curr Med Res Opin. 2006 Sep;22(9):1745-55. doi: 10.1185/030079906x120913. PMID 16968578
- [Background] Binkley N, Ringe JD, Reed JI, Ljunggren O, Holick MF, Minne HW, Liu M, Lamotta A, West JA, Santora AC. Alendronate/vitamin D3 70 mg/2800 IU with and without additional 2800 IU vitamin D3 for osteoporosis: results from the 24-week extension of a 15-week randomized, controlled trial. Bone. 2009 Apr;44(4):639-47. doi: 10.1016/j.bone.2008.05.002. Epub 2008 May 15. PMID 19185560